CLINICAL TRIAL: NCT04445584
Title: 7 Tesla MRI Evaluation of the Spine
Brief Title: 7 Tesla MRI Evaluation of the Spine (Asymptomatic)
Status: Recruiting | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Reto Sutter, MD, Chief of radiology, MD, Balgrist University Hospital
Other Study IDs: R450
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-02

CONDITIONS: Magnetic Resonance Imaging; Cervical Spine Anatomy; Reference Standard

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: 7 Tesla MRI — 7 Tesla MRI

SUMMARY:
High-resolution MRI (7 Tesla) of the cervical spine is capable to provide good differentiation between nerve and surrounding tissues within foramen und allows to reliably quantify the diameter of nerve roots/ganglia. Secondly, detailed anatomy of vertebral artery and its relation to neural structures / foramina can be assessed.

ELIGIBILITY:
Inclusion criteria:

* Informed consent as documented by signature (Appendix Informed Consent Form)
* >18 years old
* Patients presenting chronic back pain (> 2 months) without recent trauma, previous MRI (1,5 or 3T) for clinicals indications or asymptomatic individuals (for depicting normal microanatomy)

Exclusion criteria:

* previous surgery
* tumor patients
* pregnancy or breast feeding
* any MRI contra-indications
* any MRI contra-indications

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: asymptomatic individuals
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
standard values (diameter in mm) of nerve roots/ganglia/neuroforamen in each segment | 1 year
  measure the diameter of the neuroforamen (in mm) and the diameter of each cervical nerve root/ganglion within the neuroforamen (in mm)

SECONDARY OUTCOMES:
relation of vertebral artery to neural structures - assessment of contact between ganglion/spinal nerve and vertebral artery by assessing the presence of fat tissue between these structures. | 1 year
  to assess if there is contact between the vertebral artery and the ganglion/spinal nerve at each segment and each side if no fat tissue is interposed between the ganglion and vertebral artery it is classified as having contact. If contact is present, the length of contact (in mm) will be measured in the axial plane.

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No